CLINICAL TRIAL: NCT04968535
Title: Effect of Regular Electrotherapy in Patients With Chronic Non-specific Neck Pain and Low-back Pain: a Randomized Controlled Double-blinded Pilot Trial
Brief Title: Effect of Regular Electrotherapy in Patients With Chronic Non-specific Neck Pain and Low-back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Asami Naka, Sponsor-Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS-621000-0687-002
Record Dates: First submitted 2021-04-13; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Chronic Low-back Pain; Chronic Pain; Back Pain Without Radiation
Keywords: electrotherapy; chronic back pain; range of motion
MeSH Terms: conditions — Chronic Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled double blinded pilot study
Who Masked: Participant, Investigator
Masking Description: Randomization was performed using a Computer based randomization program. The physician regulating the electrotherapy device was the only one who was unmasked. The others (physician recruiting the patients, physician investigating the patients at the beginning and in the end of the enrollment, nurses) as well as the patients were blinded. The team was instructed to keep conversations to a minimum required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Therapy (Experimental): Patients receiving suprathreshold electrotherapy in weekly intervals for a Duration of 30 min each. Device calibration with determination of the individual threshold was performed prior to the application of electrical current.
  Interventions: Device: StimaWELL
- Control (Sham Comparator): Patients receiving device calibration without consequent electrotherapy.
  Interventions: Device: StimaWELL
- Control of control (No Intervention): Patients lay on the mat without receiving device calibration nor electrotherapy.

INTERVENTIONS:
Device: StimaWELL — mid frequent electrotherapy mat covering the whole spinal cord with different stimulation protocols installed
  Arms: Control; Therapy

SUMMARY:
This randomized controlled double-blinded pilot trial was performed in the Medical University of Vienna, Department of Special Anesthesia and Pain Medicine between 2015 and 2018. Aim of the study was to assess the effect of regular electrotherapy applied on the spinal cord of patients with chronic non-specific neck pain and/or low-back pain. The hypothesis was that subjective feeling of pain, range of motion of the cervical and lumbar region, as well as the activity in daily living improved after weekly electrotherapy sessions for 30 min each.

DETAILED DESCRIPTION:
Chronic neck pain and low-back pain are common causes for the decrease in quality of life. Unfortunately, efficacy of medical therapy is limited (Maher et al, 2017), and evidence for the efficacy of transcutaneous electrical nerve stimulation (TENS) therapy for both chronic neck pain (Martimbianco et al, 2019), as well as for chronic low-back pain (Khadilkar et al, 2008) is scarce .

With the aim to assess the effectiveness of regular electrotherapy in chronic pain patients applied via a mat covering the whole spinal cord, and thus allowing deeper current penetration into the tissue compared to conventional TENS, male and female patients with chronic neck pain or low back pain aged 18 years or over were enrolled in this study.

After informed consent, patients were randomly divided in three groups: Group 1 (verum) received right after device calibration suprathreshold electrotherapy on the whole back for 30 min weekly, Group 2 (Control) received device calibration without consequent electrotherapy, Group 3 (Control of Control) just lay on the mat without receiving device calibration nor electrotherapy.

Electrotherapy was applied using a mat covering the whole spinal cord called "StimaWELL". Therefore, all the patients were asked to put off the clothes and lay supine on the mat for 30 min in each session.

Primary outcome was the subjective pain sensation measured with the numeric pain rating scale (NRS). Secondary outcomes were cervical and lumbar range of motion and activities in daily living.

Data recorded before and after the sessions (i.e. NRS at rest, NRS under activity, average NRS in the last four weeks, maximum and minimum NRS, and Short-form Mc Gill Pain Questionnaire for pain sensation, measurement of the lumbar range of motion using Modified Schober and measurement of cervical range of motion using the Cervical range of Motion Device (CROM), assessment of activities in daily living using the Neck Disability Index and Rolland Morris Questionnaire) was compared in each group,respectively.

Inclusion criteria were a numeric pain rating scale (NRS) equal or more than 5 prior to study enrollment, and chronic pain in the cervical or lumbar Region longer than three month.

Exclusion criteria were pregnancy, prior experience in TENS, epilepsy, cardiac arrythmia, cardiac operation prior to study enrollment including implanted pacemaker or defibrillator, operation in the spinal cord, malignancies or infectious diseases affecting the spinal cord, severe radicular pain with acute paralysis in the extremities or an ongoing pension application.

Oral pain medication had to be unchanged at least four weeks before the study enrollment. Additional pain therapies like acupuncture, physical therapy, intravenous pain therapy or intramuscular or subcutaneous injection of pain medication were not accepted.

All patients, as well as the recruiting investigator and the physician performing the physical measurements and questionnaires were blinded.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neck pain and/or low back pain longer than 3 month
* Minimum numeric pain rating scale equal or > 5

Exclusion Criteria:

* Change in pain medication within 4 weeks prior or during the enrollment (except intake of rescue medication)
* Additional pain therapies within 4 weeks prior or during the enrollment
* Epilepsy
* Pregnancy
* Previous experience in TENS
* Cardiac arrythmia/previous cardiac operation/implanted cardiac devices
* Infection or malignancies affecting the spinal cord/previous spine operation
* Severe radicular pain with acute paralysis in the extremities
* Ongoing pension application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
change in numeric pain rating scale at 8 weeks compared to baseline | 8 weeks
  Change from baseline subjective pain sensation from 0 (no pain) to 10 (maximum pain) at 8 weeks

SECONDARY OUTCOMES:
change in cervical range of motion at 8 weeks compared to baseline | 8 weeks
  Cervical range of motion measured in degree using CROM (cervical range of motion device; the higher the number, the better the mobility).
change in lumbar range of motion at 8 weeks compared to baseline | 8 weeks
  Lumbar range of motion measured in cm using the Modified Schober Method (measurement of the skin distance 10 cm above and 5 cm below the posterior superior iliac spine during anteflexion and retroflexion, respectively. The higher the value in anteflexion, the better the mobility; the smaller the measured skin distance in retroflexion, the better the mobility).
Change in activity in daily living influenced by neck pain at 8 weeks compared to baseline | 8 weeks
  Change in the activity in daily living after 8 weeks compared to baseline using a questionnaire called "Neck Disability Index" for cervicalgia: Minimum 0 points (no disability), maximum 50 Points (severe disability); score calculation: Points examined divided 50 times 100; the higher, the more disabled in daily living due to chronic neck pain.
Change in activity in daily living influenced by low back pain at 8 weeks compared to baseline | 8 weeks
  Change in the activity in daily living after 8 weeks compared to baseline using "Rolland Morris Disability Questionnaire" for low back pain: Minimum 0 points (no disability), Maximum 24 points. The higher the score, the more disabled due to low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Sator-Katzenschlager, Prof., MD, Principal Investigator — Department of Special Anesthesia and Pain Medicine, Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Martimbianco ALC, Porfirio GJ, Pacheco RL, Torloni MR, Riera R. Transcutaneous electrical nerve stimulation (TENS) for chronic neck pain. Cochrane Database Syst Rev. 2019 Dec 12;12(12):CD011927. doi: 10.1002/14651858.CD011927.pub2. PMID 31830313
- [Background] Khadilkar A, Odebiyi DO, Brosseau L, Wells GA. Transcutaneous electrical nerve stimulation (TENS) versus placebo for chronic low-back pain. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD003008. doi: 10.1002/14651858.CD003008.pub3. PMID 18843638

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT04968535/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT04968535/ICF_001.pdf